CLINICAL TRIAL: NCT01522651
Title: A Phase 2, Proof of Concept, Randomized, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Ranolazine and Dronedarone When Given Alone and in Combination on Atrial Fibrillation Burden in Subjects With Paroxysmal Atrial Fibrillation
Brief Title: Study to Evaluate the Effect of Ranolazine and Dronedarone When Given Alone and in Combination in Patients With Paroxysmal Atrial Fibrillation
Acronym: HARMONY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-291-0102; 2011-001134-42 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ranolazine; Dronedarone; Dual Chamber Pacemakers
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ranolazine; Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Ranolazine placebo plus dronedarone placebo for 12 weeks.
  Interventions: Drug: Ranolazine placebo; Drug: Dronedarone placebo
- Ranolazine 750 mg (Experimental): Ranolazine 750 mg plus dronedarone placebo for 12 weeks.
  Interventions: Drug: Ranolazine; Drug: Dronedarone placebo
- Dronedarone 225 mg (Experimental): Ranolazine placebo plus dronedarone 225 mg for 12 weeks.
  Interventions: Drug: Dronedarone; Drug: Ranolazine placebo
- Ranolazine 750 mg + Dronedarone 225 mg (Experimental): Ranolazine 750 mg plus dronedarone 225 mg for 12 weeks.
  Interventions: Drug: Ranolazine; Drug: Dronedarone
- Ranolazine 750 mg + Dronedarone 150 mg (Experimental): Ranolazine 750 mg plus dronedarone 150 mg for 12 weeks.
  Interventions: Drug: Ranolazine; Drug: Dronedarone

INTERVENTIONS:
Drug: Ranolazine — Tablets administered orally twice daily.
  Other Names: Ranexa®
  Arms: Ranolazine 750 mg; Ranolazine 750 mg + Dronedarone 150 mg; Ranolazine 750 mg + Dronedarone 225 mg
Drug: Dronedarone — Capsule administered orally twice daily
  Arms: Dronedarone 225 mg; Ranolazine 750 mg + Dronedarone 150 mg; Ranolazine 750 mg + Dronedarone 225 mg
Drug: Ranolazine placebo — Tablets administered orally twice daily.
  Arms: Dronedarone 225 mg; Placebo
Drug: Dronedarone placebo — Capsules administered orally twice daily
  Arms: Placebo; Ranolazine 750 mg

SUMMARY:
The primary objective of this study is to evaluate the effect of ranolazine and of low-dose dronedarone when given alone and in combination at different dose levels on atrial fibrillation burden (AFB) over 12 weeks of treatment. AFB is defined as the total time a participant is in atrial tachycardia/atrial fibrillation (AT/AF) expressed as a percentage of total recording time.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females aged 18 years and older
* Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* History of PAF documented within the prior 12 months

  - Patients with PAF undergoing cardioversion greater than 4 weeks prior to Screening are eligible
* Implanted (at least 3 months prior to Screening) dual chamber programmable pacemakers with AF detection capabilities
* AFB ≥ 1% and ≤ 70% between the last clinic evaluation and Screening (minimum of 1 month observation period) and AFB ≥ 2% and ≤ 70% during the Run in period
* Sexually active females of childbearing potential must agree to utilize effective methods of contraception during heterosexual intercourse throughout the treatment period and for 14 days following discontinuation of the study medication

Key Exclusion Criteria:

Disease - specific:

* Persistent AF or Permanent AF
* History of atrial flutter or atrial tachycardia without successful ablation
* Other acutely reversible causes of AF, including but not limited to: hyperthyroidism, pericarditis, myocarditis, or pulmonary embolism
* New York Heart Association (NYHA) Class III and IV heart failure or NYHA Class II heart failure with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic within 4 weeks prior to Screening.
* Recent history of left ventricular ejection fraction (LVEF) < 40%
* Myocardial infarction, unstable angina, or coronary artery bypass graft (CABG) surgery within three months prior to Screening or percutaneous coronary intervention (PCI) within 4 weeks prior to Screening
* Clinically significant valvular disease in the opinion of the Investigator
* Stroke within 3 months prior to Screening
* History of serious ventricular arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation) within 4 weeks prior to Screening
* Family history of long QT syndrome
* Corrected QT interval (QTc) ≥ 500 msec (Bazett) at Screening ECG if in sinus rhythm (SR). If in AF, evidence of QTc ≥ 500 msec (Bazett) within 4 weeks prior to Screening
* Prior heart transplant
* Cardiac ablation within 4 months prior to Screening, or planned ablation during the course of the study

Concomitant medications/food

* Need for concomitant treatment during the trial, with drugs or products that are strong inhibitors of cytochrome P450 3A (CYP3A), or inducers of CYP3A

  - Such medications should be discontinued 5-half lives prior to the Run-in period
* Use of grapefruit juice or Seville orange juice during the study
* Use of Class I and Class III antiarrhythmic drugs other than amiodarone within 5-half lives prior to the Run-in period
* Use of amiodarone within 3 months prior to Screening
* Use of drugs that prolong the QT interval
* Previous use of ranolazine or dronedarone within 2 months prior to screening
* Prior use of ranolazine or dronedarone which was discontinued for safety or tolerability
* Use of dabigatran during the study
* Use of digitalis preparations (eg, digoxin) during the study
* Use of a greater than 1000 mg total daily dose of metformin during the study

Laboratory tests:

* Hypokalemia (serum potassium < 3.5 mEq/L) at Screening that cannot be corrected to a level of potassium ≥ 3.5 mEq/L prior to randomization
* Moderate and severe hepatic impairment (ie, Child-Pugh Class B and C), abnormal liver function test defined as alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin > 2 x upper limit of normal (ULN) at Screening
* Severe renal impairment defined as creatinine clearance ≤ 30 mL/min at Screening

Others:

* Females who are pregnant or are breastfeeding
* In the judgment of the Investigator, any clinically-significant ongoing medical condition that might jeopardize the individual's safety or interfere with the study, including participation in another clinical trial within the previous 30 days using a therapeutic modality which could have potential residual effects that might confound the results of this study
* Any device-related technical issue which in the judgment of the investigator would disrupt adequate data collection or interpretation (eg, anticipated pulse generator change or lead revision)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2014-03-10 (Actual); Study Completion 2014-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (49):
- United States (15):
  - Investigational Site, Beverly Hills, California
  - Investigational Site, Newport Beach, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Aurora, Colorado
  - Investigational Site, Washington D.C., District of Columbia
  - Investigational Site, Lakeland, Florida
  - Investigational Site, Takoma Park, Maryland
  - Investigational Site, Towson, Maryland
  - Investigational Site, Utica, New York
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Warwick, Rhode Island
  - Investigational Site, Houston, Texas
  - Investigational Site, Murray, Utah
  - Investigational Site, Seattle, Washington
  - Investigational Site, Wausau, Wisconsin
- Germany (8):
  - Investigational Site, München, Bavaria
  - Investigational Site, Würzburg, Bavaria
  - Investigational Site, Bonn, North Rhine-Westphalia
  - Investigational Site, Coburg
  - Investigational Site, Frankfurt
  - Investigational Site, Göttingen
  - Investigational Site, Ingolstadt
  - Investigational Site, Lübeck
- Israel (8):
  - Investigational Site, Ashkelon, Ashqelon
  - Investigational Site, Afula, Zefat
  - Investigational Site, Hadera
  - Investigational Site, Haifa
  - Investigational Site, Holon
  - Investigational Site, Jerusalem
  - Investigational Site, Nahariya
  - Investigational Site, Rehovot
- Italy (2):
  - Investigational Site, Como
  - Investigational Site, Florence
- Netherlands (2):
  - Investigational Site, Maastricht, Limburg
  - Investigational Site, Groningen
- Poland (13):
  - Investigational Site, Poznan, Greater Poland Voivodeship
  - Investigational Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Investigational Site, Krakow, Lesser Poland Voivodeship
  - Investigational Site, Warsaw, Masovian Voivodeship
  - Investigational Site, Bialystok, Podlaskie Voivodeship
  - Investigational Site, Gdansk, Pomeranian Voivodeship
  - Investigational Site, Sopot, Pomeranian Voivodeship
  - Investigational Site, Katowice, Silesian Voivodeship
  - Investigational Site, Zabrze, Silesian Voivodeship
  - Investigational Site, Szczecin, Zachodniop
  - Investigational Site, Lodz
  - Investigational Site, Warsaw
  - Investigational Site, Lodz, Łódź Voivodeship
- Investigational Site, London, England, United Kingdom

REFERENCES:
- [Derived] Reiffel JA, Camm AJ, Belardinelli L, Zeng D, Karwatowska-Prokopczuk E, Olmsted A, Zareba W, Rosero S, Kowey P; HARMONY Investigators. The HARMONY Trial: Combined Ranolazine and Dronedarone in the Management of Paroxysmal Atrial Fibrillation: Mechanistic and Therapeutic Synergism. Circ Arrhythm Electrophysiol. 2015 Oct;8(5):1048-56. doi: 10.1161/CIRCEP.115.002856. Epub 2015 Jul 30. PMID 26226999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany, Israel, Italy, Netherlands, Poland, and the United States. The first participant was screened on 24 January 2012. The last study visit occurred on 10 March 2014.
Pre-assignment Details: 327 participants were screened.
Groups:
- Placebo: Placebo to match ranolazine tablet orally twice daily + placebo to match dronedarone capsule orally twice daily for 12 weeks.
- Ranolazine 750 mg: Ranolazine 750 milligrams (mg) tablet orally twice daily + placebo to match dronedarone capsule orally twice daily for 12 weeks.
- Dronedarone 225 mg: Placebo to match ranolazine tablet orally twice daily + dronedarone 225 mg capsule orally twice daily for 12 weeks.
- Ranolazine 750 mg + Dronedarone 225 mg: Ranolazine 750 mg tablet orally twice daily + dronedarone 225 mg capsule orally twice daily for 12 weeks.
- Ranolazine 750 mg + Dronedarone 150 mg: Ranolazine 750 mg tablet orally twice daily + dronedarone 150 mg capsule orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg
Started | 26 | 27 | 26 | 28 | 27
Completed | 17 | 19 | 22 | 20 | 21
Not Completed | 9 | 8 | 4 | 8 | 6
Not completed — Adverse Event | 3 | 4 | 4 | 5 | 4
Not completed — Cardioversion | 1 | 0 | 0 | 0 | 0
Not completed — Device Malfunction | 0 | 1 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 1 | 0
Not completed — Participant Non-Compliance | 1 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 1 | 1 | 0 | 1 | 1
Not completed — Randomized but Never Treated | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received ≥ 1 dose of study drug (ranolazine/placebo tablets or dronedarone/placebo capsules).
Groups:
- Ranolazine 750 mg: Ranolazine 750 mg tablet orally twice daily + placebo to match dronedarone capsule orally twice daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg | Total
Number analyzed (Participants) | 26 | 26 | 26 | 27 | 26 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8.4) | 70 (10.8) | 75 (7.8) | 71 (7.1) | 73 (9.4) | 72 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 16 | 12 | 11 | 68
  Male | 13 | 10 | 10 | 15 | 15 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 3 | 1 | 6
  Not Hispanic or Latino | 22 | 25 | 26 | 24 | 25 | 122
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 26 | 26 | 26 | 27 | 25 | 130
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 5 | 4 | 8 | 4 | 2 | 23
  Israel | 5 | 6 | 1 | 6 | 6 | 24
  Italy | 0 | 0 | 0 | 1 | 0 | 1
  Netherlands | 0 | 0 | 0 | 0 | 1 | 1
  Poland | 10 | 12 | 11 | 11 | 15 | 59
  United States | 6 | 4 | 6 | 5 | 2 | 23

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation Burden (AFB) at Baseline
Description: AFB was defined as the total time a participant was in atrial tachycardia (AT)/atrial fibrillation (AF) expressed as a percentage of total recording time. Geometric mean is the mean of log-transformed AFB exponentiated.
Time Frame: Baseline
Population: The Full Analysis Set included randomized participants who received ≥ 1 dose of study drug (ranolazine, dronedarone, or placebo) and had ≥ 2 weeks (14 days) of AFB data for both the period from screening to Day 1 and following the start of treatment. Participants with available data were analyzed.
Measure: Geometric Mean (Standard Error); unit: Percentage of total recording time
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg
Number analyzed (Participants) | 18 | 18 | 23 | 20 | 22
Percentage of total recording time | 12.7 (2.21) | 10.8 (2.70) | 11.6 (2.47) | 11.7 (2.40) | 11.7 (2.04)

2. Primary Outcome: Percent Change From Baseline in Atrial Fibrillation Burden (AFB) by Week 12
Description: AFB was defined as the total time a participant was in atrial tachycardia (AT)/atrial fibrillation (AF) expressed as a percentage of total recording time. Data are presented for baseline-adjusted AFB over 12 weeks of treatment. Geometric mean is the mean of log-transformed AFB exponentiated.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg
Number analyzed (Participants) | 18 | 18 | 23 | 20 | 22
percent change | -5.9 (18.00) | -23.0 (21.17) | 3.5 (15.68) | -59.1 (10.47) | -45.5 (10.73)
Statistical Analysis 1: Comparison: Placebo vs Ranolazine 750 mg; Test type: Other — Pairwise Comparative analysis; p = 0.493, ANCOVA — An equal-slopes analysis of covariance (ANCOVA) model was fitted to log-transformed AFB over 12 weeks, with baseline AFB as the covariate. AFB values < 1% (> 99%) were set to 1% (99%) before transformation; Percentage Difference = -19.8, 95% CI 2-sided [-57.5 to 51.5], Standard Error of Mean 25.7
Statistical Analysis 2: Comparison: Placebo vs Dronedarone 225 mg; Test type: Other — Pairwise Comparative analysis; p = 0.780, ANCOVA — An equal-slopes ANCOVA model was fitted to log-transformed AFB over 12 weeks, with baseline AFB as the covariate. AFB values < 1% (> 99%) were set to 1% (99%) before transformation; Percentage Difference = 8.8, 95% CI 2-sided [-40.2 to 98.2], Standard Error of Mean 32.9
Statistical Analysis 3: Comparison: Placebo vs Ranolazine 750 mg + Dronedarone 225 mg; Test type: Other — Pairwise Comparative analysis; p = 0.008, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Percentage Difference = -57.0, 95% CI 2-sided [-76.8 to -20.1], Standard Error of Mean 13.4
Statistical Analysis 4: Comparison: Placebo vs Ranolazine 750 mg + Dronedarone 150 mg; Test type: Other — Pairwise Comparative analysis; p = 0.072, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Percentage Difference = -42.6, 95% CI 2-sided [-68.7 to 5.2], Standard Error of Mean 17.5
Statistical Analysis 5: Comparison: Ranolazine 750 mg vs Dronedarone 225 mg; Test type: Other — Pairwise Comparative analysis; p = 0.315, ANCOVA — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 6: Comparison: Ranolazine 750 mg vs Ranolazine 750 mg + Dronedarone 225 mg; Test type: Other — Pairwise Comparative analysis; p = 0.049, ANCOVA — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: Ranolazine 750 mg vs Ranolazine 750 mg + Dronedarone 150 mg; Test type: Other — Pairwise Comparative analysis; p = 0.275, ANCOVA — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 8: Comparison: Dronedarone 225 mg vs Ranolazine 750 mg + Dronedarone 225 mg; Test type: Other — Pairwise Comparative analysis; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 9: Comparison: Dronedarone 225 mg vs Ranolazine 750 mg + Dronedarone 150 mg; Test type: Other — Pairwise Comparative analysis; p = 0.028, ANCOVA — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 10: Comparison: Ranolazine 750 mg + Dronedarone 225 mg vs Ranolazine 750 mg + Dronedarone 150 mg; Test type: Other — Pairwise Comparative analysis; p = 0.334, ANCOVA — [p-value comment as in outcome 2, analysis 2]

3. Primary Outcome: Absolute Change From Baseline in AFB by Week 12
Description: AFB is defined as the total time a participant is in AT/AF expressed as a percentage of total recording time. Data are presented for baseline-adjusted AFB over 12 weeks of treatment.
Time Frame: Baseline; Week 12
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: percentage of total recording time
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg
Number analyzed (Participants) | 18 | 18 | 23 | 20 | 22
percentage of total recording time
  Baseline | 16.8 (3.66) | 17.3 (3.74) | 19.1 (4.14) | 16.8 (3.11) | 16.7 (3.52)
  Absolute Change From Baseline in AFB by Week 12 | 4.6 (3.19) | -3.1 (2.17) | 5.6 (2.65) | -4.7 (3.24) | -3.9 (3.11)

4. Secondary Outcome: Percentage of Participants Who Had ≥ 30%, ≥ 50%, or ≥ 70% Reduction From Baseline in AFB
Description: AFB was defined as the total time a participant was in AT/AF expressed as a percentage of total recording time.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg
Number analyzed (Participants) | 18 | 18 | 23 | 20 | 22
percentage of participants
  ≥ 30% Reduction From Baseline AFB | 22.2 | 50.0 | 21.7 | 45.0 | 54.5
  ≥ 50% Reduction From Baseline AFB | 16.7 | 22.2 | 13.0 | 45.0 | 54.5
  ≥ 70% Reduction From Baseline AFB | 11.1 | 16.7 | 8.7 | 45.0 | 27.3

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to the last dose date (maximum 102 days) plus 30 days
Description: The Safety Analysis Set included participants who received ≥1 dose of study drug (ranolazine/placebo tablets or dronedarone/placebo capsules).
Arm/Group | Placebo | Ranolazine 750 mg | Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 225 mg | Ranolazine 750 mg + Dronedarone 150 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26 | 7/26 | 2/26 | 5/27 | 1/26
Other Adverse Events (participants affected / at risk) | 9/26 | 15/26 | 14/26 | 12/27 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Ranolazine 750 mg (N=26) | Dronedarone 225 mg (N=26) | Ranolazine 750 mg + Dronedarone 225 mg (N=27) | Ranolazine 750 mg + Dronedarone 150 mg (N=26)
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Ranolazine 750 mg (N=26) | Dronedarone 225 mg (N=26) | Ranolazine 750 mg + Dronedarone 225 mg (N=27) | Ranolazine 750 mg + Dronedarone 150 mg (N=26)
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 4 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 1
Asthenia (General disorders) | 2 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 3 | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 3 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 1 | 2
Prothrombin time prolonged (Investigations) | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 2 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Haematoma (Vascular disorders) | 2 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years